CLINICAL TRIAL: NCT05937412
Title: A Comparative Study Between Honey and Alcohol as Topical Skin Disinfectant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS 312/2022
Record Dates: First submitted 2022-12-10; First posted 2023-07-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Disinfectant Causing Toxic Effect
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alcohol group (Active Comparator): 70% isopropyl alcohol will be topically applied and spread uniformly on a prespecified area of at least 3 cm x 3cm on the dorsum of the hand. A skin swab will be obtained from the selected skin area just before and 20 seconds after topical application of alcohol and honey.
  Interventions: Other: Alcohol sterilization
- honey group (Active Comparator): honey will be topically applied and spread uniformly on a prespecified area of at least 3 cm x 3cm on the dorsum of the hand. A skin swab will be obtained from the selected skin area just before and 20 seconds after topical application of alcohol and honey.
  Interventions: Other: Honey sterilization

INTERVENTIONS:
Other: Alcohol sterilization — Sterilizing skin using alcohol
  Arms: alcohol group
Other: Honey sterilization — Sterilizing skin using honey
  Arms: honey group

SUMMARY:
Skin antisepsis is essential in every healthcare environment. Alcohol/chlorhexidine use might disrupt skin microbiota and lead to antibiotic resistance.

This study investigates honey (being natural product with many beneficial therapeutic effects) as topical skin anti-septic agent and compares it with alcohol, in terms of effectiveness and safety.

DETAILED DESCRIPTION:
Recent years' investigations of the co-evolution and functional integration of the human body and its commensal microbiota have disclosed that the microbiome has a major impact on physiological functions including protection against infections.

Invasive procedures such as injections, punctures or surgeries penetrate the skin's natural protective barrier, which may allow pathogenic microorganisms to enter deeper skin layers and cavities and trigger infections there.

Alcohols usually in the form of 70% isopropyl alcohol or 60 to 80% ethyl alcohol, are commonly used topical disinfectants.

Despite being efficiently broad-spectrum antiseptic, Alcohol shows some local hazards affecting skin integrity and microbiome.

Honey has been used in wound care since ancient. It has many beneficial therapeutic effects, including anti-microbia, antioxidant, immune-modulator, wound healing and synbiotic effects .

Antimicrobial agents are important in reducing the burden of infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* - Children aged from 2 to 12 years, of both sexes, and with apparently healthy skin.
* Children, who did not receive any form of antimicrobial agent for at least one-week prior study.

Exclusion Criteria:

* - Immuno-compromised due to diseases or drugs.
* - Children having any skin disease as eczema or others

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy of honey as a disinfectant in comparison to the standard disinfectant which is alcohol | 3 months
  taking a swab from skin for culture of organisms after application of either alcohol or honey and compare type of organisms and number of colony forming units

CONTACTS AND LOCATIONS:
Overall Officials: mamdouh abdelmaksoud, Study Director — Ain Shams University; yosra awad, Study Director — Ain Shams University; maha ahmad, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breasted JH. (1930): The Edwin Smith papyrus: published in facsimile and hieroglyphic transliteration. Chicago: University of Chicago Press.
- [Background] Wiemken TL. Skin antiseptics in healthcare facilities: is a targeted approach necessary? BMC Public Health. 2019 Aug 22;19(1):1158. doi: 10.1186/s12889-019-7507-5. PMID 31438910
- [Background] Gheldof N, Engeseth NJ. Antioxidant capacity of honeys from various floral sources based on the determination of oxygen radical absorbance capacity and inhibition of in vitro lipoprotein oxidation in human serum samples. J Agric Food Chem. 2002 May 8;50(10):3050-5. doi: 10.1021/jf0114637. PMID 11982440
- [Background] Hasyimi W, Widanarni W, Yuhana M. Growth Performance and Intestinal Microbiota Diversity in Pacific White Shrimp Litopenaeus vannamei Fed with a Probiotic Bacterium, Honey Prebiotic, and Synbiotic. Curr Microbiol. 2020 Oct;77(10):2982-2990. doi: 10.1007/s00284-020-02117-w. Epub 2020 Jul 18. PMID 32683466
- [Background] Held E, Mygind K, Wolff C, Gyntelberg F, Agner T. Prevention of work related skin problems: an intervention study in wet work employees. Occup Environ Med. 2002 Aug;59(8):556-61. doi: 10.1136/oem.59.8.556. PMID 12151613
- [Background] Jull AB, Cullum N, Dumville JC, Westby MJ, Deshpande S, Walker N. Honey as a topical treatment for wounds. Cochrane Database Syst Rev. 2015 Mar 6;2015(3):CD005083. doi: 10.1002/14651858.CD005083.pub4. PMID 25742878
- [Background] Majtan J. Honey: an immunomodulator in wound healing. Wound Repair Regen. 2014 Mar-Apr;22(2):187-92. doi: 10.1111/wrr.12117. Epub 2014 Feb 24. PMID 24612472
- [Background] Mandal MD, Mandal S. Honey: its medicinal property and antibacterial activity. Asian Pac J Trop Biomed. 2011 Apr;1(2):154-60. doi: 10.1016/S2221-1691(11)60016-6. PMID 23569748
- [Background] Christensen GJ, Bruggemann H. Bacterial skin commensals and their role as host guardians. Benef Microbes. 2014 Jun 1;5(2):201-15. doi: 10.3920/BM2012.0062. PMID 24322878
- [Background] Sato T, Miyata G. The nutraceutical benefit, part iii: honey. Nutrition. 2000 Jun;16(6):468-9. doi: 10.1016/s0899-9007(00)00271-9. No abstract available. PMID 10869910
- [Background] Trevisanato SI. Treatments for burns in the London Medical Papyrus show the first seven biblical plagues of Egypt are coherent with Santorini's volcanic fallout. Med Hypotheses. 2006;66(1):193-6. doi: 10.1016/j.mehy.2005.08.052. Epub 2005 Oct 14. PMID 16226847